CLINICAL TRIAL: NCT03631264
Title: The Effect of Kinesiotaping Method on Feeding of Late Preterm Infants.
Acronym: kinesiotape
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nilay Comuk Balci, Associate Professor, Baskent University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA18/36
Record Dates: First submitted 2018-08-12; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Preterm Infants
Keywords: preterm infants; kinesiotape; swallowing
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape (Experimental): Kinesiotape application to masseter and hyoid muscles of late preterm infants for improving sucking and swallowing.
  Interventions: Device: Kinesiotape
- Control (No Intervention): In this group the late preterm infants won't be applied kinesiotaping to suck and swallow muscles.

INTERVENTIONS:
Device: Kinesiotape — Kinesiotape application to masseter and hyoid muscles of late preterm infants to improve sucking and swallowing.
  Other Names: Control
  Arms: Kinesiotape

SUMMARY:
Problems such as poor nutrition, weak sucking, lack of suck-swallow-respiration coordination, low weight gain are among the factors increasing the risk of morbidity in late preterm infants. Early support of sucking and swallowing muscles for the development of suck-swallow coordination can shorten the maturation process and provide early discharge of late preterm infants. The aim of this study is to document kinesiotape technique to support sucking and swallowing muscles for treating nutritional problems and for reducing nutrition risks and accelerating maturation. According to power of analysis of this study, 74 infants planned to assign to kinesiotaping group or control group randomly. In kinesiotaping group, infants feeding performance will be evaluated by measuring the amount of milk invested, maximum heart rate, oxygen saturation, speed of milk intake and counting the number of swallow during feeding. Kinesiotape will be applied to masseter and hyoid muscles 24 hours later after the birth of the infant. Infants will be evaluated before kinesiotape application, 3 hour later and 24 hour later after the application.

ELIGIBILITY:
Inclusion Criteria:

* Infants born in Baskent University Ankara Hospital, age between 34-36.6 weeks.

Exclusion Criteria:

* Infants with multiple kongenital anomaly, hypoxic ischemic encephalopathy, intraventricular and intracranial hemorrhage, necrotizing enterocolitis, tracheoesophageal fistula, diaphragmatic hernia, hydrocephalus, and respiratory distress.

Ages: 34 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
digital stethoscope | 2 minutes
  It helps to count the number of swallows of the baby during feeding

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Anuk Ince, MD, Study Director — Associate Professor
Locations (1):
- Baskent University Ankara Hospital, Ankara, Bahçelievler, Turkey (Türkiye)